CLINICAL TRIAL: NCT02032953
Title: Enhancing the Anabolic Effect of Perioperative Nutrition With Insulin While Maintaining Normoglycemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Thomas Schricker, Chief of Anesthesia, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-459-GEN
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; protein recovery; perioperative nutrition; hyperinsulinemia; normoglycemia; hyperinsulinemic-normoglycemic clamp; anabolism
MeSH Terms: conditions — Colorectal Neoplasms; Hyperinsulinism | interventions — amino-acid, glucose, and electrolyte solution; Amino Acids; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Insulin, Travasol (35%) postop (Experimental): Insulin (hyperinsulinemic-normoglycemic clamp) with Travasol (amino acid supplementation) given from start of surgery to 6 hours after, at an amount of 35% of patient's energy expenditure as measured before surgery, .
  Interventions: Dietary Supplement: Travasol (amino acid injection); Drug: Insulin
- Insulin, Travasol (20%) postop (Experimental): Insulin (hyperinsulinemic-normoglycemic clamp) with Travasol (amino acid infusion), given from start of surgery to 6 hours after, at an amount of 20% of patient's energy expenditure as measured before surgery.
  Interventions: Dietary Supplement: Travasol (amino acid injection); Drug: Insulin
- Insulin, no protein after surgery (Placebo Comparator): Insulin (hyperinsulinemic-normoglycemic clamp, an insulin infusion between 2 and 5 microunits/kg with glucose at a variable rated titrated to maintain normoglycemia, blood glucose 4-6 mmol/L) with no protein supplementation from start of surgery to 6 hours after.
  Interventions: Drug: Insulin

INTERVENTIONS:
Dietary Supplement: Travasol (amino acid injection) — an amino acid supplementation infused intravenously containing essential and non-essential amino acids
  Other Names: Travasol
  Arms: Insulin, Travasol (20%) postop; Insulin, Travasol (35%) postop
Drug: Insulin — After the insertion of an arterial catheter and obtaining a baseline arterial blood glucose value, 2 units of insluin will be administered iv followed by an infusion of 2 microunits/kg*min. Ten minuts after starting the insulin, and when the the blood glucose is<6 mmol/L, dextrose 20% supplemented with phosphate (30mmol/L) will be infused. Blood glucose levels measured every 15 minutes and the dextrose infusion rate adjusted to maintain arterial glycemia between 4 and 6 mmol/L until end of study.
  Other Names: HNC; Hyperinsulinemic-normoglycemic clamp

SUMMARY:
The purpose of this study is to find out whether adding insulin after current colorectal cancer surgery promotes making and keeping proteins in the body, and to find out whether or not this effect can be further increased by increasing the amount of protein given.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class<3
* age>18 years
* colorectal surgery for non-metastatic colorectal adenocarcinoma including right and left hemicolectomy, transverse, subtotal and total colectomy sigmoid and low anterior resection
* ability to give informed consent

Exclusion Criteria:

* BMI>30 Kg/meter squared
* confirmed diagnosis of diabetes mellitus or a HbA1c>6.0%
* significant cardiorespiratory, hepatic, renal and neurological disease
* musculoskeletal or neuromuscular disease
* ingestion of drugs known to affect protein, glucose and lipid metabolism (e.g. steroids)
* severe anemia (hemoglobin<10 g/dL
* pregnancy
* history of severe sciatica, back surgery or other conditions which contraindicate the use of epidural catheters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-12; Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Net protein balance | 6 hours after surgery
  The difference in total body protein after randomization to one of the three treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schricker, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre (MUHC) - Royal Victoria Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Schricker T, Meterissian S, Wykes L, Eberhart L, Lattermann R, Carli F. Postoperative protein sparing with epidural analgesia and hypocaloric dextrose. Ann Surg. 2004 Nov;240(5):916-21. doi: 10.1097/01.sla.0000143249.93856.66. PMID 15492576
- [Result] Schricker T, Wykes L, Carli F. Epidural blockade improves substrate utilization after surgery. Am J Physiol Endocrinol Metab. 2000 Sep;279(3):E646-53. doi: 10.1152/ajpendo.2000.279.3.E646. PMID 10950834
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194